CLINICAL TRIAL: NCT06177470
Title: Effectiveness of Accelerated Transcranial Magnetic Stimulation in Obsessive Compulsive
Brief Title: Effectiveness of Accelerated Deep TMS in OCD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Selim Tumkaya, Professor, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023TIPF023
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: obsessive compulsive disorder; intermittant Teta Burst Transcranial Magnetic Stimulation; accelerated TMS; Transcranial Magnetic Stimulation
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active accelerated deep TMS (Active Comparator): Accelerated dTMS on anterior cingulate cortex and medial prefrontal cortex.
  Interventions: Device: Accelerated deep iTBS
- sham TMS (Sham Comparator): Sham TMS on anterior cingulate cortex and medial prefrontal cortex
  Interventions: Device: Accelerated Sham iTBS

INTERVENTIONS:
Device: Accelerated deep iTBS — Accelerated intermittant teta burst deep Transcranial Magnetic Stimulation on anterior cingulate cortex and medial prefrontal cortex 50 Hz
  Arms: active accelerated deep TMS
Device: Accelerated Sham iTBS — Sham accelerated intermittant teta burst Transcranial Magnetic Stimulation on anterior cingulate cortex and medial prefrontal cortex 50 Hz
  Arms: sham TMS

SUMMARY:
H-coil high-frequency deep transcranial magnetic stimulation (dTMS) over the medial prefrontal cortex (mPFC) and anterior cingulate cortex (ACC) has been approved by the Food and Drug Administration for use in treatment-resistant obsessive-compulsive disorder. At the same time, there are studies in the literature showing the effectiveness of intermittent theta burst stimulation application and the advantages of short treatment duration. However, there is no strong scientific evidence yet on the effectiveness and safety of iTBS (50 Hz) application with a double-cone coil in obsessive-compulsive disorder patients. The aim of this study is to evaluate the effectiveness of dTMS with ITBS protocol on the medial prefrontal cortex (mPFC) and anterior cingulate cortex (ACC) in OCD patients.

DETAILED DESCRIPTION:
The current study aimed to investigate the effectiveness and safety of the ITBS protocol, which is applied to the mPFC and ACC for 5 sessions per day with a double-cone coil in treatment-resistant OCD patients. This study evaluated (I) the effectiveness of Itbs (50 Hz) stimulation of the mPFC and ACC with a double-cone coil and (II) the effectiveness of administering this protocol over 2 weeks rather than six weeks as approved by the FDA. Participants will be randomized into two parallel groups in a double-blind manner. In one group, ITBS (50 Hz) dTMS will be applied to mPFC and ACC, and in the other group, sham tms will be applied to the same regions. The application consists of a total of 50 sessions, 5 times a day. This application will last for a total of 10 days excluding weekends.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of obsessive-compulsive disorder
* Not having an adequate response to treatment despite the use of an SGI selective serotonin reuptake inhibitors at a sufficient dose and duration (at least 8 weeks) before the planned add-on treatment
* No dose or active substance changes have been made in the treatment regimen for at least 8 weeks
* Aged 18-65 years
* Able to read and write
* Not having a significant medical or neurological disease

Exclusion Criteria:

* Not providing consent to participate in the study
* Diagnosis of a psychiatric disorder, such as psychotic disorder, bipolar disorder, major depressive disorder [Hamilton Depression Rating Scale (HDRS) score above 17], mental retardation, alcohol-substance use disorder, and organic mental disorder (dementia, delirium, and head trauma, etc.)
* Diagnosis of an important medical or neurological disease (e.g., epilepsy);
* Mental retardation
* Illiteracy
* Having received electroconvulsive therapy (ECT) or TMS within the last six months;
* Having any prosthesis, such as an implant and pacemaker.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-18 (Estimated); Primary Completion 2024-09-18 (Estimated); Study Completion 2024-10-18 (Estimated)

PRIMARY OUTCOMES:
Obsessive compulsive symptoms severity | pretreatment (0.days) - as soon as the work is completed (10. days) - In the 2nd week after TMS application is completed (24. days)
  Yale-Brown Obsessive-Compulsive Scale (Y-BOCS). The minimum and maximum values are 0-40, and higher scores mean a worse outcome.
Dimensional obsessive compulsive symptom severity | pretreatment (0.days) - as soon as the work is completed (10. days) - In the 2nd week after TMS application is completed (24. days)
  Dimensional Obsessive-Compulsive Scale (DOCS). The minimum and maximum values are 0-80, and higher scores mean a worse outcome.

SECONDARY OUTCOMES:
Severity of Depression | pretreatment (0.days) - as soon as the work is completed (10. days) - In the 2nd week after TMS application is completed (24. days)
  Hamilton Depression Rating Scale. The minimum and maximum values are 0-52, and higher scores mean a worse outcome
Severity of anxiety | pretreatment (0.days) - as soon as the work is completed (10. days) - In the 2nd week after TMS application is completed (24. days)
  Hamilton Anxiety Rating Scale. The minimum and maximum values are 0-56, and higher scores mean a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Selim Tümkaya, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cole EJ, Stimpson KH, Bentzley BS, Gulser M, Cherian K, Tischler C, Nejad R, Pankow H, Choi E, Aaron H, Espil FM, Pannu J, Xiao X, Duvio D, Solvason HB, Hawkins J, Guerra A, Jo B, Raj KS, Phillips AL, Barmak F, Bishop JH, Coetzee JP, DeBattista C, Keller J, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Accelerated Intelligent Neuromodulation Therapy for Treatment-Resistant Depression. Am J Psychiatry. 2020 Aug 1;177(8):716-726. doi: 10.1176/appi.ajp.2019.19070720. Epub 2020 Apr 7. PMID 32252538
- [Background] Cole EJ, Phillips AL, Bentzley BS, Stimpson KH, Nejad R, Barmak F, Veerapal C, Khan N, Cherian K, Felber E, Brown R, Choi E, King S, Pankow H, Bishop JH, Azeez A, Coetzee J, Rapier R, Odenwald N, Carreon D, Hawkins J, Chang M, Keller J, Raj K, DeBattista C, Jo B, Espil FM, Schatzberg AF, Sudheimer KD, Williams NR. Stanford Neuromodulation Therapy (SNT): A Double-Blind Randomized Controlled Trial. Am J Psychiatry. 2022 Feb;179(2):132-141. doi: 10.1176/appi.ajp.2021.20101429. Epub 2021 Oct 29. PMID 34711062
- [Background] Carmi L, Tendler A, Bystritsky A, Hollander E, Blumberger DM, Daskalakis J, Ward H, Lapidus K, Goodman W, Casuto L, Feifel D, Barnea-Ygael N, Roth Y, Zangen A, Zohar J. Efficacy and Safety of Deep Transcranial Magnetic Stimulation for Obsessive-Compulsive Disorder: A Prospective Multicenter Randomized Double-Blind Placebo-Controlled Trial. Am J Psychiatry. 2019 Nov 1;176(11):931-938. doi: 10.1176/appi.ajp.2019.18101180. Epub 2019 May 21. PMID 31109199
- [Background] Carmi L, Alyagon U, Barnea-Ygael N, Zohar J, Dar R, Zangen A. Clinical and electrophysiological outcomes of deep TMS over the medial prefrontal and anterior cingulate cortices in OCD patients. Brain Stimul. 2018 Jan-Feb;11(1):158-165. doi: 10.1016/j.brs.2017.09.004. Epub 2017 Sep 6. PMID 28927961
- [Derived] Akyol GK, Yucens B, Tumkaya S. Accelerated deep intermittent theta-burst stimulation for obsessive-compulsive disorder: A double-blind, randomized, controlled study. J Psychiatr Res. 2025 Sep;189:365-372. doi: 10.1016/j.jpsychires.2025.06.034. Epub 2025 Jun 24. PMID 40578057